CLINICAL TRIAL: NCT04033471
Title: Effect of Epidural Morphine and Midazolam on Postoperative Painin Patients Undergoing Major Abdominal Cancer Surgery
Brief Title: Combined Epidural Morphine and Midazolam on Postoperative Pain
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Shereen Mamdouh, associate professor of anesthesia, ICU and pain manegement, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 464
Record Dates: First submitted 2019-07-24; First posted 2019-07-26 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Acute Postoperative Pain
Keywords: epidural, morphine, midazolam, acute postoperative pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Midazolam; Morphine; Bupivacaine

STUDY DESIGN:
Intervention Model Description: epidural bupiviacain
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MI (Active Comparator): Bupivacaine 0.25% + midazolam 5mg in total volume 10m1
  Interventions: Drug: midazolam
- MM (Active Comparator): Bupivacaine 0.25% + midazolam 5mg and morphine 5mg in total volume 10ml
  Interventions: Drug: midazolam
- MO (Active Comparator): bupivacaine 0.25% + morphine 5 mg in total volume 10 ml
  Interventions: Drug: midazolam

INTERVENTIONS:
Drug: midazolam — epidural needle in the L1-2 or L2-3 space , and using loss of resistance technique udder strict aseptic condition 10 ml of the prepared drug will be given
  Other Names: morphine; bupivacaine

SUMMARY:
this study aim to Compare the effect of preoperative Epidural Midazolam, Morphine and their combination in postoperative pain relief and total morphine consumption.

DETAILED DESCRIPTION:
Major abdominal surgeries with abdominal incisions lead to severe abdominal pain, which if treated inadequately, can cause shallow breathing, atelectasis, retention of secretions and lack of cooperation in physiotherapy. This increases the incidence of post-operative morbidity and leads to delayed recovery.Epidural anesthesia is safe and inexpensive technique with the advantage of providing surgical anesthesia and prolonged postoperative pain relief. It also an effective treatment of operative pain blunts autonomic, somatic and endocrine responses. Morphine and midazolam can be used as adjuvant to bupivicain to reduced the postoperative pain

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II patients scheduled for major abdominal cancer surgeries

Exclusion Criteria:

* patients with known allergy to the study drugs,
* significant cardiac, respiratory, renal or hepatic disease,
* drug or alcohol abuse,
* psychiatric illness that would interfere with perception and assessment of pain.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2021-03 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
time to first request of analgesia | 1st 48 hours postoperative
  the time between the end of operation and tracheal extubation to the first request for supplemental analgesics and its administration to the patient

SECONDARY OUTCOMES:
the cumulative consumption of morphine in the 1st 48h postoperatively | 1st 48 hours postoperative
  total amount of morphine used for analgesia

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt